CLINICAL TRIAL: NCT03794245
Title: Bringing South African Men Into HIV Counseling (HCT) and Care
Brief Title: Bringing South African Men Into HIV Counseling and Testing and Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Human Sciences Research Council (Other Government); Medical University of South Carolina (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Thomas J. Coates, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH105534 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2019-01-04 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: Prevention; Testing and Diagnosis; Treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Disease

STUDY DESIGN:
Intervention Model Description: Men-Centered HIV Testing vs. Clinic-Based HIV Testing; Personalized Linkage to Care for HIV+ Men vs. Clinic Referral for HIV+ Men.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The Care Provider and Outcomes Assessors do not know the arms to which an individual has been assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Men-Centered HIV Testing (Experimental): Mobile HIV testing is conducted at sites in the community where men gather.
  Interventions: Behavioral: Men-Centered HIV Testing
- Clinic-based HIV Testing (Active Comparator): Men are referred to the nearest clinic for HIV counseling and testing
  Interventions: Behavioral: Clinic-based HIV Testing
- Linkage to Care for HIV+ Men (Experimental): The patient coordinator arranges an appointment time at the clinic and accompanies the patient to the initial visit
  Interventions: Behavioral: Linkage to Care for HIV+ Men
- Clinic Referral for HIV+ Men (Active Comparator): Men diagnosed with HIV are referred to the nearest clinic for treatment of HIV
  Interventions: Behavioral: Clinic Referral for HIV+ Men

INTERVENTIONS:
Behavioral: Men-Centered HIV Testing — The intervention involves bringing mobile HIV testing to venues where men congregate, talking to them as a group about HIV testing, and then providing testing at that venue.
  Arms: Men-Centered HIV Testing
Behavioral: Linkage to Care for HIV+ Men — Men diagnosed with HIV are accompanied to the clinic and registered there with the help of a community health worker.
  Arms: Linkage to Care for HIV+ Men
Behavioral: Clinic-based HIV Testing — Individuals present to a clinic and request HIV counseling and testing
  Arms: Clinic-based HIV Testing
Behavioral: Clinic Referral for HIV+ Men — Individuals diagnosed with HIV are referred to the nearest clinic for treatment of HIV
  Arms: Clinic Referral for HIV+ Men

SUMMARY:
This clinical trial seeks to determine if male-centered recruitment increases men's testing for HIV and whether or not individualized introduction to clinics increases male engagement in treatment for HIV. The study is being conducted in rural KwaZulu Natal.

DETAILED DESCRIPTION:
This study combines structural and individual level interventions for HIV and integrates the two to address the study's objective of identifying South African men in KwaZulu Natal with HIV and maintaining those diagnosed with HIV in care to the point of viral suppression.

The cluster-randomized design will randomize 8 communities to intervention or control to test the hypothesis whether male-centered mobilization and testing increases the population-level percentage of men who have been tested within the past 12 months by more than 10 absolute percentage points.

The individually randomized design will test whether individualized case management will effectively link HIV-positive men to treatment to the point of viral suppression.

The study will also examine the incremental cost-effectiveness of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Men residing in the target communities

Exclusion Criteria:

* Men outside of the target communities
* Men who report being tested and HIV+

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1806 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of men tested for HIV | Tested within the past 12 months
  Percentage of men in the community, selected through probability sampling, who report being tested for HIV

OTHER OUTCOMES:
Percentage of HIV+ men initiating treatment for HIV | Within 6 months of receiving HIV diagnosis
  Percentage of men HIV+ enrolling in treatment centers and starting treatment for HIV
Percentage of men with suppressed viral load | 12 months after initiating treatment
  Percentage of men with HIV viral load <50 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: THOMAS J COATES, PhD, Principal Investigator — University of California, Los Angeles; Heidi Van Rooyen, PhD, Principal Investigator — Human Sciences Research Council
Locations (1):
- Human Sciences Research Council, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Rooyen H, Makusha T, Joseph P, Ngubane T, Kulich M, Sweat M, Coates T. Zwakala Ndoda: a cluster and individually randomized trial aimed at improving testing, linkage, and adherence to treatment for hard-to reach men in KwaZulu-Natal, South Africa. Trials. 2019 Dec 30;20(1):798. doi: 10.1186/s13063-019-3908-0. PMID 31888701